CLINICAL TRIAL: NCT01138982
Title: A Randomized Effectiveness Trial of a One-to-one, Adult-to-youth Mentoring Program in Sweden
Brief Title: Effectiveness Study of a Swedish Youth Mentoring Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Ministry of Health and Social Affairs, Sweden (Other Government); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Maria Bodin, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dnr 238/2006:34
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Substance Use
Keywords: Youth mentoring; Effectiveness; Sweden; low-risk youth
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mentoring program (Experimental): Mentor and mentee meet at least every second week, for 2-4 h on every occasion, during 1 year (i.e., for a minimum of two school semesters). Meetings take place outside school and work hours, and the pairs choose activities of their own preferences. No monetary incentives exist, and the mentors are laymen volunteers. The program objective is to establish a safe and supportive relationship, by which the youth is assumed to benefit in social, emotional, and academic development, and as a consequence, be less prone to use alcohol and drugs.
  Interventions: Behavioral: Youth Mentoring program
- Control group (No Intervention): No intervention provided, only brief phone calls to control for attention bias

INTERVENTIONS:
Behavioral: Youth Mentoring program
  Arms: Mentoring program

SUMMARY:
This study aims to investigate the effectiveness of a one-to-one, adult-to-youth primary preventive mentoring program in Sweden. Outcome domains and criteria for inclusion and exclusion of study participants are elaborated in collaboration with the providing NGO, and the program is given as customary.

ELIGIBILITY:
Inclusion Criteria:

* a self-reported need of the youth for additional adult contacts

Exclusion Criteria:

* current or past regular use of illicit drugs
* repeated delinquent behaviour or single acts of violence against persons
* ongoing contacts with psychiatric care or social services

Ages: 14 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Self-reported substance use | One year
  Self-reported substance use among youth

SECONDARY OUTCOMES:
Youth delinquency | One year
  Self-reported delinquency among youth

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Bodin, PhD, Principal Investigator — Centre for Psychiatry Research Stockholm, Karolinska Institutet/Stockholm County Council Health Care Provision
Locations (1):
- Mentor Sweden, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No